CLINICAL TRIAL: NCT02154503
Title: Evaluating the Efficacy of Microneedling in the Treatment of Androgenetic Alopecia- Pilot Study
Brief Title: Evaluating the Efficacy of Microneedling in the Treatment of Androgenetic Alopecia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vancouver General Hospital (Other)
Responsible Party: Principal Investigator, Jerry Shapiro, Clinical Professor, Vancouver General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H13-03501
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Microneedling (Experimental): By randomization, the side for treatment will be determined. Topical anaesthetic will be then placed onto the treatment area under occlusion for thirty minutes to one hour. This will then be removed with 70% alcohol. The area will be rolled with microneedles in two planes: coronally and sagitally. In each plane, five passes will be made. Patients will restart application of Minoxidil the following day to both sides of the lesion.
  The same half of the scalp will be treated for the rest of the sessions, with topical anaesthetic applied by patient 30 minutes to an hour prior to start of treatment session. Patients will undergo microneedling on alternate weeks for a total of six treatments in 12 weeks. If there is >30% growth seen after six weeks, then the entire area will be treated.
  Interventions: Device: topical 5% Minoxidil (Microneedling)

INTERVENTIONS:
Device: topical 5% Minoxidil (Microneedling)

SUMMARY:
Androgenetic Alopecia is the most common non scarring alopecia worldwide. Treatment of which has been limited with few options for medical and surgical treatment, the cost of the latter being prohibitive for many. Recently there have been several new modalities proposed as treatment, namely Microneedling and Platelet Rich Plasma.

Microneedling has been shown to overexpress hair growth factors which may enhance or stimulate miniaturized hairs to grow. It has also been shown to increase the absorption of topical products significantly. The exact mechanism of action of Microneedling is still being delineated.

In this study, we aim to do a half lesional study with global photographs and hair counts done at the start of , week four and week twelve. Patients would be needled once weekly after application of topical anaesthetic (5% EMLA). If by week six there is significant regrowth (>30%), then total lesional needling will be done. Patients will only be using topical 5% Minoxidil throughout the study as this will prolong the effects of the regrowth.

ELIGIBILITY:
Inclusion Criteria:

1. Men between the ages 18-65.
2. Disease Stage: Norwood Hamilton IIIa-IV.
3. Length of time with disease < 10 years.

Exclusion Criteria:

1. Must not have other concurrent hair disease.
2. Have not used any oral anti androgen (Finasteride or Dutasteride) in the past six months. If so, a washout period is needed. One month for Finasteride and three months for Dutasteride.
3. Patients under the age of 18.
4. Patients who are unable to offer consent.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Hair caliber diameter and hair counts will be measured on both the treated and untreated sides. | three months

SECONDARY OUTCOMES:
Adverse effects of the procedure will be recorded. | three months

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Shapiro, MBBS, Principal Investigator — University of British Columbia
Locations (1):
- The Skin Care Centre, Vancouver, British Columbia, Canada